CLINICAL TRIAL: NCT07148167
Title: Cervical MRI Findings in Patients With Ankylosing Spondylitis
Brief Title: Comparison of Cervical Extensor Muscle Thickness, Fat Infiltration, and Cervical Alignment in Patients With Ankylosing Spondylitis With a Healthy Population: a Retrospective Controlled Study
Status: Completed | Type: Observational
Sponsor: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Guc, Medical Doctor, Kayseri City Hospital
Other Study IDs: Kayseri City EAH
Record Dates: First submitted 2025-07-14; First posted 2025-08-29 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-05

CONDITIONS: Muscle Planes, Muscle Volumes, Fat Infiltration in Cervical MRI
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ankylosing Spondylitis group: For the study group:
  * Patients diagnosed with ankylosing spondylitis, aged 18-50.
  * Patients who underwent a cervical MRI between January 2020 and September 2023.
  Interventions: Other: Magnetic resonance imaging
- Control Group: Patients aged 18-50 who underwent cervical MRI between January 2020 and September 2023 due to nonspecific neck pain, who did not have an AS diagnosis and whose cervical MRI was reported as normal.
  Interventions: Other: Magnetic resonance imaging

INTERVENTIONS:
Other: Magnetic resonance imaging — use Magnetic Resonance Imaging (MRI) to evaluate the cervical muscle planes in AS patients in more detailed and objective ways. In this study, in addition to cervical muscle volumes in AS patients, we also aimed to evaluate cervical fat infiltration and cervical alignment, which have not been previously evaluated in AS patients.

SUMMARY:
In the literature, we found only one study evaluating the thickness of the cervical paraspinal muscles (multifidus, semispinalis cervicis, semispinalis capitis, splenius capitis, and trapezius) in patients with AS. This study examined the morphology of all neck extensor muscles (multifidus, semispinalis capitis, semispinalis cervicis, splenius capitis, and trapezius muscles) using ultrasound and their relationship to activities of daily living and compared them with a control group. As is well known, the user's experience is crucial in ultrasound. Furthermore, ultrasound cannot accurately assess the deep paravertebral muscles. Therefore, inspired by this study, we decided to use Magnetic Resonance Imaging (MRI) to evaluate the cervical muscle planes in AS patients in more detailed and objective ways. In this study, in addition to cervical muscle volumes in AS patients, we also aimed to evaluate cervical fat infiltration and cervical alignment, which have not been previously evaluated in AS patients.

ELIGIBILITY:
Inclusion Criteria:

* For the study group:
* Patients diagnosed with ankylosing spondylitis, aged 18-50.
* Patients who underwent a cervical MRI between January 2020 and September 2023. Control Group Patients aged 18-50 who underwent cervical MRI between January 2020 and September 2023 due to nonspecific neck pain, who did not have an AS diagnosis and whose cervical MRI was reported as normal.

Exclusion Criteria:

* Patients over 50 years of age
* History of spine surgery;
* Presence of pain, numbness, and weakness in the upper extremities
* History of cervical injury or neck injury
* Presence of tuberculosis, tumor, fracture, infection, instability, cervical myelopathy, cervical disc herniation (protrusion, extrusion) (will be considered cervical bulging)
* Presence of cervical radiculopathy
* Those with a detectable pathological spinal condition related to neck pain, including spinal deformity; inflammatory or rheumatic diseases other than AS, malignancies, or neurological diseases
* A cognitive or psychological disorder

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: For the study group:
  * Patients diagnosed with ankylosing spondylitis, aged 18-50.
  * Patients who underwent a cervical MRI between January 2020 and September 2023. Control Group Patients aged 18-50 who underwent cervical MRI between January 2020 and September 2023 due to nonspecific neck pain, who did not have an AS diagnosis and whose cervical MRI was reported as normal.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
servical MRI fındings in AS patients, | Patients who underwent cervical MRI between January 2020 and September 2023
  the cervical muscle planes, cervical muscle volumes in AS patients cervical fat infiltration

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri City Hospital, Kayseri, Kocasinan, Turkey (Türkiye)